CLINICAL TRIAL: NCT05808283
Title: Preoperative Anemia Frequency
Status: Completed | Type: Observational
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Gamze Küçükosman, medical doctor, Zonguldak Bulent Ecevit University
Other Study IDs: 2021/20
Record Dates: First submitted 2023-03-29; First posted 2023-04-11 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Preoperative Evaluation
Keywords: preoperative evaluation; preoperative anemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Those with anemia according to WHO definition (Group 1)
  Interventions: Other: preoperative anemia frequency
- Those without anemia according to WHO definition (Group 2)
  Interventions: Other: preoperative anemia frequency

INTERVENTIONS:
Other: preoperative anemia frequency — patients who applied to the outpatient clinic prospectively for 3 months
  Other Names: blood transfusion frequency

SUMMARY:
In our retrospective study, it was aimed to determine the frequency of anemia in non-emergency patients over the age of 18 who applied to the Anesthesiology and Reanimation Department of our hospital.

ELIGIBILITY:
Inclusion Criteria:

* -patient over 18 years old,
* Patients applying to the Department of Anesthesiology and Reanimation AD

Exclusion Criteria:

* Pregnant,
* under 18 years old,
* will undergo cardiac and emergency surgery
* Patients with Massive Bleeding
* Patients who underwent multiple surgeries during the study period

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years of age, without massive bleeding, of both sexes
Sampling Method: Non-Probability Sample
Enrollment: 853 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
PREOPERATIVE ANEMIA FREQUENCY AND TREATMENT APPROACH | Patients who applied to the outpatient clinic within a 3-month period after ethical approval
  preoperative anemia frequency

SECONDARY OUTCOMES:
PREOPERATIVE ANEMIA FREQUENCY AND TREATMENT APPROACH | Patients who applied to the outpatient clinic within a 3-month period after ethical approval
  blood transfusion frequency

CONTACTS AND LOCATIONS:
Locations (1):
- Gamze Küçükosman, Zonguldak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided